CLINICAL TRIAL: NCT03910179
Title: Dynamic Arterial Elastance as Predictive Parameter of Hypotension During General Anesthesia Induction.
Brief Title: Dynamic Arterial Elastance During General Anesthesia Induction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Professor, Università Politecnica delle Marche
Other Study IDs: CLRIA-AC01
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates if dynamic arterial elastance measured before general anesthesia induction can predict the occurrence of hypotension due to general anesthesia induction.

DETAILED DESCRIPTION:
As general anesthetics may be responsible for vasodilation and cardiac depression, arterial hypotension after induction of general anesthesia is a common event and may contribute to an adverse outcome. Dynamic arterial elastance has been proposed as a functional parameter of arterial tone and studies showed that it was able to predict pressure response to fluid administration in fluid-responsive patients and the amount of mean arterial pressure riduction as a conseguence of noradrenaline dose reduction in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will be undergone to general anesthesia for surgery
* Patients that need mini-invasive cardiac output monitoring during surgery

Exclusion Criteria:

* Age <18 yo
* Pregnancy
* Arrhythmia
* Severe valvular diseases
* Uncorrectable alterations of arterial signal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone to general anesthesia for surgery that need mini-invasive cardiac output monitoring.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Baseline value of Eadyn as predictor of hypotension occurrence due to general anesthesia induction | From baseline (before general anesthesia induction) up to 30 minutes.
  Dynamic arterial elastance (Eadyn) will be recorded at baseline before induction of general anesthesia. Mean arterial pressure (MAP) will be recorded at baseline and continuously until tracheal intubation. The lowest value of MAP will be considered to define hypotension occurrence.

SECONDARY OUTCOMES:
Correlation between Eadyn and severity of hypotension due to anesthesia induction | From baseline (before general anesthesia induction) up to 30 minutes.
  To evaluate the correlation between the baseline value of Eadyn and the severity of hypotension when it will occur after induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, PhD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- Azienda ospedaliero Universitaria Ospedali Riuniti Ancona, Ancona, Italy